CLINICAL TRIAL: NCT02689570
Title: Relation of Visceral Fat and Associated Cytokines With Early Cardiovascular Complications in Type 1 Diabetes: the VISCERA Study
Brief Title: Relation of Visceral Fat and Associated Cytokines With Early Cardiovascular Complications in Type 1 Diabetes.
Acronym: VISCERA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Antwerp (Other)
Collaborators: Universiteit Antwerpen (Other)
Responsible Party: Principal Investigator, Christophe De Block, MD PhD, University Hospital, Antwerp
Other Study IDs: VISCERA
Record Dates: First submitted 2016-02-11; First posted 2016-02-24 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-02

CONDITIONS: Type 1 Diabetes; Coronary Artery Calcifications; Diastolic Dysfunction
Keywords: type 1 diabetes; coronary artery calcifications; diastolic dysfunction; adipokines; visceral adipose tissue
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Watchful Waiting; Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — EDTA sample
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- type 1 diabetic patients: Adult T1DM patients, aged 18-75 years, regularly attending the out-patient diabetes clinic of the Antwerp University Hospital are recruited starting from June 2011. Patients had to have a diabetes duration of ≥5 years and be in general good health to be included. Exclusion criteria were a history of a major adverse cardiovascular event (myocardial infarction, stroke), other cardiovascular complaints, pregnancy or a glomerular filtration rate ≤30 ml/min/1.73 m2.
  Interventions: Other: observational

INTERVENTIONS:
Other: observational — no interventions; observational study
  Other Names: no interventions; observational study

SUMMARY:
Objective: To investigate whether visceral adipose tissue (VAT) and its adipokines contribute to early signs of cardiovascular disease, meaning coronary artery calcifications (CAC) and diastolic dysfunction in type 1 diabetes (T1DM).

Research Design & Methods: A cross-sectional study of T1DM patients without a history of cardiovascular disease. CAC and VAT are measured using a CT scan. CAC is scored using the Agatston method. Echocardiography is performed to assess contractile abnormalities. Serum levels of adipocytokines (adiponectin, leptin, IL-6 and TNF-a) are measured using ELISA assays.

DETAILED DESCRIPTION:
Objective: To investigate whether visceral adipose tissue (VAT) and its adipokines contribute to early signs of cardiovascular disease, meaning coronary artery calcifications (CAC) and diastolic dysfunction in type 1 diabetes (T1DM).

Patients & Methods:

Adult T1DM patients, aged 18-75 years, regularly attending the out-patient diabetes clinic of the Antwerp University Hospital are recruited starting from June 2011. Patients have to have a diabetes duration of ≥5 years and be in general good health to be included. Exclusion criteria are a history of a major adverse cardiovascular event (myocardial infarction, stroke), other cardiovascular complaints, pregnancy or a glomerular filtration rate ≤30 ml/min/1.73 m².

All participants sign an informed consent form. This study is conducted in accordance with the amended Declaration of Helsinki. The research protocol is approved by the Antwerp University Hospital Ethics committee (UZA 11/31/224, Belgian registration number: B30020111874).

Anthropometric measurements:

All measurements are performed in the morning after an overnight fast. Height is measured to the nearest 0.5 cm using a wall-mounted stadiometer, and weight is measured using a balance beam scale with subjects in their underwear. Waist circumference is measured at the mid-level between the lower rib margin and the iliac crest. Body composition is assessed by bio-impedance analysis (BIA) and fat mass percentage is calculated using the formula of Deurenberg. Visceral abdominal adipose tissue (VAT) and subcutaneous abdominal adipose tissue (SAT) are determined by a 64-slice computerized tomography (CT) scan at the L4-L5 level (slice thickness 0.6mm).

Blood pressure is taken with a standardized method (Dynamap) after a 10-min rest, and a mean of four measurements is used. Hypertension is defined as blood pressure ≥130/85 mmHg or antihypertensive medication intake by the patient.

Presence of the metabolic syndrome is evaluated using the International Diabetes Federation criteria. Subjects are classified as having the metabolic syndrome if ≥3 of the following criteria are met: (1) increased waist circumference (men ≥94 cm, women ≥80 cm), (2) hypertriglyceridemia (≥150 mg/dl=1.7 mmol/l), (3) low HDL cholesterol (<40 mg/dl=1.03 mmol/l in men and <50 mg/dl=1.29 mmol/l in women), (4) high blood pressure (≥130/85 mmHg), (5) high fasting glucose (≥100 mg/dl).

Insulin resistance is determined using the inverse of the estimated glucose disposal rate (eGDR), calculated using the formula: : eGDR= 21.158 + (- 0.09 * waist circumference) + (- 3.407 * hypertension) + (- 0.551 * HbA1c).

Laboratory measurements:

HbA1C is determined by high performance liquid chromatography on an Adams™ A1c HA-8160 8180 , Arkray - Menarini instrument (Zaventem, Belgium; reference range: 4.8-6.0%). A mean of four annual determinations of A1C is used to assess overall metabolic control over the past two years. Plasma Serum levels of creatinin, total cholesterol, HDL cholesterol and triglycerides are measured on a Vitros 750 XRC (Ortho Clinical Diagnostic, Johnson & Johnson, Buckinghamshire, UK) Dimension Vista 1500 System (Siemens Healthcare Diagnostics, Huizingen, Belgium) with reagents from the same manufacturer (REF K1270A for creatinin, REF K1027 for total cholesterol, REF K3048A for HDL-cholesterol, REF K2069 for triglycerides). HDL-C is measured on a Hitachi 912 (Roche Diagnostics, Mannheim, Germany). Serum creatinine is measured by an enzymatic method on a Vitros 750 (Ortho Clinical Diagnostic, Beerse, Belgium). The glomerular filtration rate (eGFR) is estimated using the abbreviated MDRD formula, including a correction factor of 0.742 for women. Plasma HMW adiponectin concentrations are measured by an enzyme-linked immunosorbent assay (ELISA) (EZHMWA-64K, Millipore, analytical sensitivity 0.5 ng/ml, intra-assay coefficient of variation [CV] 7.47%). Leptin is measured using an ELISA kit (HU Leptin kit, KAC2281, Life Technologies, sensitivity 3.5 pg/ml, intra-assay CV 5.75%). TNF-α is assayed using ELISA (HU TNF alpha kit, KHC3011, Life Technologies, sensitivity 1.7 pg/ml, intra-assay CV 6.38%) and IL-6 concentrations are measured using ELISA (HU IL-6 Chemiluminescence Elisa kit, KHC0069, Life Technologies, sensitivity 0.25 pg/ml, intra-assay CV 5.37%).

Assessment of complications:

Each subject is assessed for presence and severity of complications. 24h-Urinary albumin is measured by nephelometry Dimension Vista 1500 System (Siemens Healthcare Diagnostics, Huizingen, Belgium) with reagents from the same manufacturer (REF K7062). using a Behring Nephelometer II (Siemens Healthcare Diagnostics Products, Marburg, Germany). Microalbuminuria is defined as a urinary albumin excretion exceeding 20 µg/min. Both carotid arteries are examined using a carotid duplex scanner (General Electrics, Vivid 7 Pro), equipped with an 8-Mhz high-resolution probe.

A 64-slice non-contrast multidetector CT scan of the coronary arteries is performed to measure coronary artery calcifications (CAC) (Lightspeed, VCT; General Electric Medical Systems, Waukesha, Wis, Milwaukee, USA). Scoring is done by one skilled radiologist (R. Salgado), who is blinded to the subjects case files. Typical imaging parameters are: tube voltage 100 kv; current intensity 310 mA; rotation time 500 ms; and detector collimation 64 x 0.625 mm. Scan data are reconstructed at 75% of the cardiac cycle after the QRS complex. The radiation dose for calcium scoring range at 1.3-1.7 mSv. CAC is quantified (Agatston score) by means of a dedicated software application (SmartScore, AW). The Agatston score is the product of CAC area times the density. A score <10 is considered as normal. A score >200 is a strong predictor of CVD risk.

Standard 2-dimensional and Doppler Echocardiography (iE-33 Philips, The Netherlands) is performed by a single cardiologist blinded to the clinical status of the study participants. Briefly, left ventricular function is assessed by the parasternal long axis M-mode and modified biplane Simpson method. Diastolic function is determined taking into account all the following parameters: mitral inflow, pulmonary vein inflow signal and mitral annular tissue Doppler (tD) velocities from end expiratory cycles according to the ASE recommendations.

ELIGIBILITY:
Inclusion Criteria:

* type 1 diabetic patients (criteria for diagnosis by the American Diabetes Association
* diabetes duration ≥5 years
* general good health

Exclusion Criteria:

* having experienced a major adverse cardiovascular event (myocardial infarction,stroke)
* having cardiovascular complaints
* pregnancy
* having an estimated glomerular filtration ≤ 30ml/min/1.73 m²

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult type 1 diabetic patients regularly attending the out-patient diabetes clinic of the Antwerp University Hospital
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2011-06; Primary Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
coronary artery calcifications | once at the moment of inclusion of this cross-sectional, observational study
  A 64-slice non-contrast multidetector CT scan of the coronary arteries was performed to measure coronary artery calcifications (CAC) (Lightspeed, VCT; General Electric Medical Systems, Waukesha, Wis, Milwaukee, USA). Scoring was done by one skilled radiologist (R. Salgado), who was blinded to the subjects case files. Typical imaging parameters were: tube voltage 100 kv; current intensity 310 mA; rotation time 500 ms; and detector collimation 64 x 0.625 mm. Scan data were reconstructed at 75% of the cardiac cycle after the QRS complex. The radiation dose for calcium scoring ranged at 1.3-1.7 mSv. CAC was quantified (Agatston score) by means of a dedicated software application (SmartScore, AW). The Agatston score is the product of CAC area times the density.

SECONDARY OUTCOMES:
diastolic dysfunction | once at the moment of inclusion of this cross-sectional, observational study
  Standard 2-dimensional and Doppler Echocardiography (iE-33 Philips, The Netherlands) was performed by a single cardiologist blinded to the clinical status of the study participants. Briefly, left ventricular function was assessed by the parasternal long axis M-mode and modified biplane Simpson method. Diastolic function was determined taking into account all the following parameters: mitral inflow, pulmonary vein inflow signal and mitral annular tissue Doppler (tD) velocities from end expiratory cycles

CONTACTS AND LOCATIONS:
Overall Officials: Luc F Van Gaal, MD, PhD, Principal Investigator — Universiteit Antwerpen
Locations (1):
- Antwerp University Hospital, Edegem, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] De Block CEM, Shivalkar B, Goovaerts W, Brits T, Carpentier K, Verrijken A, Van Hoof V, Parizel PM, Vrints C, Van Gaal LF. Coronary artery calcifications and diastolic dysfunction versus visceral fat area in type 1 diabetes: VISCERA study. J Diabetes Complications. 2018 Mar;32(3):271-278. doi: 10.1016/j.jdiacomp.2017.11.008. Epub 2017 Nov 28. PMID 29310998